CLINICAL TRIAL: NCT00377390
Title: Inner-City Anti-IgE Therapy for Asthma Mechanistic Study
Brief Title: ICATA Asthma Mechanistic Study
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: DAIT ICAC-09
Record Dates: First submitted 2006-09-14; First posted 2006-09-18 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2013-02

CONDITIONS: Asthma
Keywords: Immunoglobulin; IgE; Omalizumab
MeSH Terms: conditions — Asthma | interventions — Omalizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples, sputum, and nasal secretions

GROUPS / COHORTS (2):
- Cockroach sensitive
  Interventions: Biological: Omalizumab
- Control (cockroach insensitive)
  Interventions: Biological: Omalizumab

INTERVENTIONS:
Biological: Omalizumab — Subcutaneous injections of omalizumab will be administered every 2 or 4 weeks along with standardized asthma care for 60 weeks, beginning with the Randomization Visit, as a part of ICATA (ICAC-08, NCTNCT00377572).

SUMMARY:
The purposes of this study are to determine the effects of omalizumab on cells involved in the allergic response, to evaluate predictors of response to omalizumab, and to determine whether response to omalizumab therapy is influenced by the environment. A subset of inner-city children and adolescents currently enrolled in Inner-City Anti-IgE Therapy for Asthma (a clinical trial of omalizumab) will be enrolled in this study.

DETAILED DESCRIPTION:
Immunoglobulin E (IgE) is important in the development of allergic responses and may determine asthma severity. Omalizumab is a man-made monoclonal antibody that directly blocks the cause of allergic reactions. There are three main objectives to this study. The first is to gain an understanding of how omalizumab affects cells involved in the immune response. The second objective is to determine whether response to omalizumab is influenced by exposure to environmental factors, including allergens and viral infections. The third objective is to determine what clinical markers can be used to determine which patients would most benefit from omalizumab therapy. This study will evaluate the immune and allergic responses of inner-city children with moderate to severe asthma who are receiving omalizumab or placebo as part of a parallel study (Inner-City Anti-IgE Therapy for Asthma, ICAC-08, NCT00377572).

Nasal secretions will be collected from all participants at the beginning of this study, toward the middle of the study, and with each asthma exacerbation requiring a clinical visit. Some participants will participate in either the basophil or T-cell studies and associated procedures. These studies require blood collection at five study visits. Sputum collection will occur at four study visits. Those participants involved in the basophil studies will also undergo skin testing at three study visits.

ELIGIBILITY:
Inclusion Criteria:

* Currently enrolled in ICATA (ICAC-08, NCT00377572) Clinical Study
* Positive skin test to German cockroach required for participation in the basophil and T-cell studies and associated procedures
* Cockroach insensitive participants will serve as control groups

Ages: 6 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Inner-city children and adolescents ages 6 to 20 with asthma who are currently enrolled in the ICATA Clinical Study
Sampling Method: Non-Probability Sample
Enrollment: 224 (Actual)
Dates: Start 2006-10; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Correlation of changes in basophil receptor occupancy with a reduction in maximum symptom days, inhaled corticosteroid dosage, sputum, and peripheral blood eosinophils, and frequency of exacerbations | 1.5 years

SECONDARY OUTCOMES:
Effect of omalizumab therapy on basophil activation markers | 1.5 years
Effect of omalizumab therapy on the skin test response to allergen and correlation of this change in skin test endpoint titration with maximum symptom days | 1.5 years
Effect of omalizumab therapy on the skin test response to allergen and correlation of this change in skin test endpoint titration with inhaled corticosteroid dosage, sputum and peripheral blood eosinophils, and frequency of exacerbations | 1.5 years

CONTACTS AND LOCATIONS:
Overall Officials: William W. Busse, MD, Study Chair — University of Wisconsin, Madison; Jacqueline Pongracic, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago; Carolyn Kercsmar, MD, Principal Investigator — Rainbow Babies and Children's Hospital; Rebecca S. Gruchalla, MD, PhD, Principal Investigator — University of Texas Southwestern Medical Center; Hugh Sampson, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (4):
- United States (4):
  - Children's Memorial Hospital, Chicago, Illinois
  - Mount Sinai School of Medicine, New York, New York
  - Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - University of Texas Southwestern Medical Center, Dallas, Texas

REFERENCES:
- [Background] Courtney AU, McCarter DF, Pollart SM. Childhood asthma: treatment update. Am Fam Physician. 2005 May 15;71(10):1959-68. PMID 15926412
- [Background] Federico MJ, Liu AH. Overcoming childhood asthma disparities of the inner-city poor. Pediatr Clin North Am. 2003 Jun;50(3):655-75, vii. doi: 10.1016/s0031-3955(03)00045-2. PMID 12877240
- [Background] Mvula M, Larzelere M, Kraus M, Moisiewicz K, Morgan C, Pierce S, Post R, Nash T, Moore C. Prevalence of asthma and asthma-like symptoms in inner-city schoolchildren. J Asthma. 2005 Feb;42(1):9-16. doi: 10.1081/jas-200044746. PMID 15801322
- [Background] Szefler SJ, Apter A. Advances in pediatric and adult asthma. J Allergy Clin Immunol. 2005 Mar;115(3):470-7. doi: 10.1016/j.jaci.2004.12.1123. PMID 15753890
- See also: Click here for more information on DAIT ICAC-08 — http://clinicaltrials.gov/ct/show/NCT00377572